CLINICAL TRIAL: NCT03426098
Title: A Prospective, Single-center, Investigator-blinded Trial to Evaluate the Safety and Efficacy of Secret Micro-Needle Fractional RF System® for the Treatment of Facial Wrinkles
Brief Title: Secret Micro-Needle Fractional RF System® for the Treatment of Facial Wrinkles
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Goldman, Butterwick, Fitzpatrick and Groff (Other)
Collaborators: Ilooda Co., Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0922-1228
Record Dates: First submitted 2018-02-02; First posted 2018-02-08 (Actual); Last update posted 2019-05-10 (Actual); Status verified 2019-05

CONDITIONS: Aging; Wrinkle

STUDY DESIGN:
Intervention Model Description: All subjects will receive up to three treatments at four week intervals to their full faces with the Secret RF device.
Masking Description: Blinded-investigator assessments will be performed at Baseline and Days 28, 56, 146, and 180 to evaluate treatment efficacy for facial wrinkling. Of note, the blinded-investigators will be blinded to treatment settings and technique, and number of treatments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Treatment (Experimental): After baseline evaluation, all subjects will undergo a series of 3 facial treatments with the Secret Micro-Needle Fractional RF System® at 4 week intervals.
  Interventions: Device: Secret RF

INTERVENTIONS:
Device: Secret RF — A series of 3 facial treatments with the Secret Micro-Needle Fractional RF System® at 4 week intervals.

SUMMARY:
To assess the safety, efficacy and patient satisfaction associated with the treatment of facial wrinkles using the Secret Micro-Needle Fractional RF System® (Ilooda Co., Ltd., Suwon, South Korea).

DETAILED DESCRIPTION:
Subjects satisfying all inclusion and exclusion criteria will be enrolled in this trial. After baseline evaluation, all subjects will undergo a series of 3 facial treatments with the Secret Micro-Needle Fractional RF System® at 4 week intervals.

Blinded-investigator and subject self-assessments will be performed at Baseline and Days 28, 56, 146, and 180 to evaluate treatment efficacy for facial wrinkling. Of note, the blinded-investigators will be blinded to treatment settings and technique, and number of treatments. Safety will be evaluated by subject diaries, as well as investigator- and subject-rated evaluations of adverse events at all follow-up visits. Mandatory standard 2D digital photography, Canfield VISIA and VECTRA 3D digital photography will be performed at baseline and at each office visit.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females in good general health who are greater than 22 years of age.
2. Subjects may be of Fitzpatrick Skin Types I through VI.
3. Subjects must desire improvement of facial skin texture and wrinkling.
4. Subjects must have at least a score of 2 on the Fitzpatrick Wrinkle Scale evaluating the forehead, cheeks, and periorbital areas and Modified Fitzpatrick Wrinkle Scale evaluating the nasolabial folds (Appendix A1 and A2).
5. Subjects must be willing to provide written informed consent, HIPAA authorization, and photographic release.
6. Subjects must be willing to follow study instructions and complete all required visits.
7. Negative urine pregnancy test results at the time of study entry (if applicable).
8. The subject is healthy as judged by medical history and investigator's assessment of current health
9. Female subjects will be either of non-childbearing potential defined as:

1. Having no uterus. 2. No menses for at least 12 months. Or; (WOCBP) women of childbearing potential must agree to use an effective method of birth control during the course of the study, such as:

1. Oral contraceptive pill, injection, implant, patch, vaginal ring, intrauterine device (systemic birth control must have been started 30 days or more prior to enrolling)
2. Intrauterine coil
3. Bilateral tubal ligation
4. Barrier method used with an additional form of contraception (e.g., sponge, spermicide or condom)
5. Abstinence (If practicing abstinence must agree to use barrier method described above (4) if becomes sexually active).
6. Vasectomized partner (Must agree to use barrier method described above (4) if becomes sexually active with non-vasectomized).

Exclusion Criteria:

1. A subject who has undergone treatment with any non-ablative laser, including IPL, within the last 3 months and any ablative laser within the last 6 months.
2. A subject who has undergone any microneedling treatment within the last 3 months
3. A subject with a history of previous fat transfer, injectable calcium hydroxylapatite or poly-l-lactic acid to the study area within the past 6 months.
4. A subject with a history of injection of hyaluronic acid dermal fillers in the study area within the past six months.
5. Retinoid, hydroquinone, microdermabrasion, or chemical peel treatments to the face within one month prior to study participation or during the study.
6. Current participation or participation within 30 days prior to the start of this study in a drug or other investigational research studies.
7. Presence of an active systemic or local skin disease that may affect wound healing.
8. Presence of scarring, sunburn, tattoos, open wounds or other skin condition in area to be treated that would interfere with the assessments of this study.
9. Individuals who have current skin cancers or suspicious lesions in the treatment area per Investigator.
10. Individuals who are nursing, pregnant, or planning to become pregnant during the study.
11. Patients who have a history with keloid formation or hypertrophic scarring.
12. Inability to understand the protocol or to give informed consent.
13. Subjects with deep dermal scarring or thick sebaceous skin of the treatment area.
14. History of impaired immune system, including but not limited to HIV, current malignancy.
15. History of chronic drug or alcohol abuse.
16. Current smoker or history of smoking in the last one year.
17. Subjects with known bleeding disorder or is receiving medication that will likely increase the risk of bleeding as the result of injection per investigator discretion.
18. Concurrent therapy that, in the investigator's opinion, would interfere with the evaluation of the safety or efficacy of the study device.
19. Subjects who anticipate the need for surgery or overnight hospitalization during the study.
20. Subjects who, in the investigator's opinion, have a history of poor cooperation, noncompliance with medical treatment, or unreliability.
21. History of using the following prescription medications:

    1. Current use of psychiatric drugs that in the investigators opinion would impair the subject from understanding the protocol requirements or understanding and signing the informed consent.
    2. Immunosuppressive medications.
22. Subjects with implantable cardiac devices, such as pacemakers or implantable cardioverter-defibrillators.

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-02-10 (Actual); Primary Completion 2019-05-30 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
Wrinkles | Baseline to Day 146
  Improvement in Wrinkles Based on the Fitzpatrick Wrinkle Scale

SECONDARY OUTCOMES:
Rating of Non-Sequential Images | Baseline, Day 28, and Day 56.
  Ratings of non-sequential images of subjects at baseline, Day 28, and Day 56. Improvement is defined as a minimum improvement by a score of 1 on the Fitzpatrick Wrinkle Scale or Modified Fitzpatrick Wrinkle Scale as graded by two out of three blinded evaluators, who will be blinded to treatment settings and technique, and number of treatments
Global Aesthetic Improvement Score | Baseline to Day 28, 56, and 146
  Investigator Assessed Global Aesthetic Improvement Score
Subject Satisfaction | Baseline to Day 28, 56, and 146
  Subject-assessed Satisfaction with Facial Appearance scale (FACE-Q)

CONTACTS AND LOCATIONS:
Overall Officials: Mitchel P Goldman, MD, Principal Investigator — Cosmetic Laser Dermatology and West Dermatology Research
Locations (1):
- West Dermatology Research Center, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No